CLINICAL TRIAL: NCT06089668
Title: A Prospective Observational Study to Evaluate Clinical Characteristics, Current Practice and Outcomes of Adult Patients With Suspected or Confirmed Melioidosis
Brief Title: An Observational Study to Evaluate Clinical Characteristics of Adult Patients With Suspected or Confirmed Melioidosis
Status: Completed | Type: Observational
Sponsor: AN2 Therapeutics, Inc (Industry)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: MEL-OB1
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Melioidosis
Keywords: Melioidosis
MeSH Terms: conditions — Melioidosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational Study — None, this is a non-interventional trial

SUMMARY:
This is a prospective observational study to evaluate clinical characteristics, current practice and outcomes of adult patients (age ≥18 years) with suspected or confirmed melioidosis.

DETAILED DESCRIPTION:
This is a prospective observational study to evaluate clinical characteristics, current practice and outcomes of adult patients (age ≥18 years) with suspected or confirmed melioidosis. Determination of microbiologically confirmed acute melioidosis among patients presenting with suspected melioidosis, and determination of clinical outcomes of interest (including all-cause mortality, characterization of organ involvement or organ failure, resolution of sepsis, improvement of renal function, rates of suspected vs. microbiologically confirmed melioidosis, and rates of melioidosis involvement of different organ systems) will be performed. Defining clinical and microbiological outcomes in a standardized manner will enable characterization and selection of the relevant outcome measures to be utilized in future clinical studies of IV epetraborole in acute melioidosis. Patients will be identified through daily, active surveillance of hospital admissions at the investigative sites and review of microbiology laboratory culture results. Data will be extracted from hospital and outpatient medical charts. These data will refine the expected treatment effect of standard-of-care antimicrobial therapy and the consequent statistical power calculations needed for sample size and outcome measure design elements of future clinical trials of IV epetraborole adjunctive therapy in hospitalized patients with suspected acute melioidosis.

Participation in the study requires written informed consent from the patient or from their next-of-kin (if needed) at the time of screening. On day 28 (+7) and day 90 (+7) after enrolment the study team will contact the participant by phone interview with standardized script if the participant is discharged alive prior to the day 28 or day 90. There will be no clinical specimens collected as part of the study protocol, as this study aims to observe clinical characteristics and outcomes among patients with confirmed and suspected acute melioidosis in current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years old and greater.
2. Thai and Laos nationality (for study site in Thailand and Laos, respectively).
3. Required hospitalization
4. Community-acquired infection is suspected as the cause of illness (Related terms - e.g. fever, acute fever, community-acquired sepsis, and other infectious diseases [e.g. r/o infectious disease, r/o malaria, r/o dengue, r/o bacteraemia and r/o leptospirosis])

For melioidosis-suspected group ONLY 4a. Community-acquired infection is suspected as the cause of illness (Related terms - e.g. fever, acute fever, community-acquired sepsis, and r/o other infectious diseases [e.g. r/o infectious disease, r/o malaria, r/o dengue, r/o bacteraemia and r/o leptospirosis]) 5a. Hospitalized (at study hospital) for less than 24 hours 6a. Suspected of melioidosis (at least one of the following)

* Ceftazidime or Meropenem has already been prescribed BEFORE screening
* SEPTIC SHOCK (sepsis at screening is defined as SOFA≥2 or qSOFA≥1; and shock at screening is defined as requiring vasopressor to maintain MAP≥65 mmHg)
* SEPSIS (defined as SOFA≥2 or qSOFA≥1) with AN UNDERLYING DISEASE of diabetes, chronic kidney disease, major thalassemia, cancer or on immunosuppressive drug (including steroid)

For melioidosis-confirmed group ONLY 4b. Have any specimen culture or Immunofluorescence Microscopy (IFM) or Polymerase Chain Reaction (PCR) positive for B. pseudomallei 5b. Patient is still in the study hospital (i.e. alive) on the screening day

Exclusion Criteria:

For Melioidosis-suspected Group ONLY

1. Have confirmed diagnosis of other infectious diseases (e.g. malaria, dengue, leptospirosis) at screening based on rapid diagnostic tests or confirmatory diagnostic tests
2. Non-infectious disease (e.g. stroke, heart attack) is suspected to be a primary cause of the sepsis or shock
3. Hospital-acquired infection is suspected by attending physician as the cause of illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Thailand and Laos with suspected or confirmed melioidosis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Data Collection of patients in Thailand with "suspected melioidosis" | 2 years
  Describe, prospective data collection, the presenting clinical characteristics of patients hospitalized in Thailand with "suspected melioidosis" to understand the presentation of this disease in a contemporaneous, rigorously studied cohort.
Data Collection of patients in Thailand with "microbiologically confirmed melioidosis ". | 2 years
  Describe, prospective data collection, the presenting clinical characteristics of patients hospitalized in Thailand with "microbiologically confirmed melioidosis " to understand the presentation of this disease in a contemporaneous, rigorously studied cohort.
Data Collection of patients in Laos with "suspected melioidosis" | 2 years
  Describe, prospective data collection, the presenting clinical characteristics of patients hospitalized in Laos with "suspected melioidosis" to understand the presentation of this disease in a contemporaneous, rigorously studied cohort.
Data Collection of patients in Laos with "microbiologically confirmed melioidosis ". | 2 years
  Describe, prospective data collection, the presenting clinical characteristics of patients hospitalized in Laos with "microbiologically confirmed melioidosis " to understand the presentation of this disease in a contemporaneous, rigorously studied cohort.

SECONDARY OUTCOMES:
Use ± Immunofluorescence Microscopy (IFM) to Determine the percentage of "suspected melioidosis patients" with microbiologically confirmed disease | 2 Years
  Use ± IFM to determine the percentage of "suspected melioidosis patients" with microbiologically confirmed disease
Use ± Polymerase Chain Reaction (PCR) to Determine the percentage of "suspected melioidosis patients" with microbiologically confirmed disease | 2 Years
  Use ± PCR to determine the percentage of "suspected melioidosis patients" with microbiologically confirmed disease
Determine the rates of Burkholderia pseudomallei eradication in patients with microbiologically confirmed acute melioidosis | 28 days after enrollment
  Determine microbiological eradication patients with microbiologically confirmed acute melioidosis
Determine frequency of specific involvement of organ systems involvement in patients with microbiologically confirmed acute melioidosis | 28 days after enrollment
  Determine the frequency of specific organ system involvement in patients with microbiologically confirmed acute melioidosis
Measure rate to resolution of bacteremia conversion to negative cultures | 28 days after enrollment
  Microbiological outcomes in patients with microbiologically confirmed acute melioidosis
Measure time to resolution of bacteremia conversion to negative cultures | 28 days after enrollment
  Microbiological outcomes in patients with microbiologically confirmed acute melioidosis
Frequency of Liver involvement in patients with microbiologically confirmed acute melioidosis (as diagnosed per standard of care) | 28 days after enrollment
  Frequency of involvement of organ systems in patients with microbiologically confirmed acute melioidosis
Frequency of Skin involvement in patients with microbiologically confirmed acute melioidosis (as diagnosed per standard of care) | 28 days after enrollment
  Frequency of involvement of organ systems in patients with microbiologically confirmed acute melioidosis
Frequency of Lung involvement in patients with microbiologically confirmed acute melioidosis (as diagnosed per standard of care) | 28 days after enrollment
  Frequency of involvement of organ systems in patients with microbiologically confirmed acute melioidosis
Frequency of Spleen involvement in patients with microbiologically confirmed acute melioidosis (as diagnosed per standard of care) | 28 days after enrollment
  Frequency of involvement of organ systems in patients with microbiologically confirmed acute melioidosis
Time to resolution of sepsis | enrollment through day 90
  Time in days to resolution of sepsis in patients with microbiologically confirmed acute melioidosis who receive antimicrobial therapy directed against B. pseudomallei
Time to resolution of fever | enrollment through day 90
  Time in days to resolution of fever in patients with microbiologically confirmed acute melioidosis who receive antimicrobial therapy directed against B. pseudomallei
Time to resolution of hypotension | enrollment through day 90
  Time in days to resolution of hypotension in patients with microbiologically confirmed acute melioidosis who receive antimicrobial therapy directed against B. pseudomallei
Determine clinical cure rates among patients with of microbiologically confirmed acute melioidosis who are treated with ceftazidime | enrollment through day 90
  Percentage of each clinical outcome of microbiologically confirmed acute melioidosis by antimicrobial treatment regimen
Determine clinical cure rates among patients with microbiologically confirmed acute melioidosis who are treated with meropenem | enrollment through day 90
  Percentage of each clinical outcome of microbiologically confirmed acute melioidosis by antimicrobial treatment regimen
Determine clinical cure rates among patients with suspected melioidosis who are treated with an appropriate antibiotic in the subset of patients with no other microbiologically confirmed diagnosis | enrollment through day 90
  Percentage of each clinical outcome of "suspected melioidosis patients" to an appropriate antibiotic (ceftazidime or meropenem) in the subset of patients with no other microbiologically confirmed diagnosis (monomicrobial acute melioidosis)
Antimicrobial durations of treatment of microbiologically confirmed acute melioidosis | enrollment through day 90
  Antimicrobial durations of treatment of microbiologically confirmed acute melioidosis (including parenteral therapy during the initial phase of treatment and oral therapy during the eradication phase)

CONTACTS AND LOCATIONS:
Locations (3):
- Mahosot Hospital, Vientiane, Laos
- Thailand (2):
  - Srinagarind Hospital, Khon Kaen
  - Sunpasitthiprasong Hospital, Ubon Ratchathani